CLINICAL TRIAL: NCT03311061
Title: Evaluation of Curriculum for Teen Pregnancy Prevention: Decisions, Responsibility, Empowerment, Accountability, Motivations & Success (DREAMS) in Houston TX
Brief Title: Evaluation of Curriculum for Teen Pregnancy Prevention: Decisions, Responsibility, Empowerment, Accountability, Motivations & Success
Acronym: DREAMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Winter Rose Services, LLC (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dawn Marie Baletka, CEO, Winter Rose Services, LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00004955
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Teen Pregnancy
Keywords: Teen Pregnancy; Prevention; Positive Youth Development; Financial Literacy; College and Career Readiness; School Based Intervention; Age 13-19; Behavior Modification

STUDY DESIGN:
Intervention Model Description: Two groups of participants. group A will receive the DREAMS Curriculum intervention. Group B (Control group) will receive curriculum already in place at school.
Who Masked: Participant
Masking Description: Students are masked through
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DREAMS (Experimental): The experimental group will be exposed to the DREAMS curriculum including the supplemental technology based application.It is composed of 10 modules: Introduction; Self Exploration; Healthy Relationships; Adolescent Sexuality; Attitudes and Adolescent Sexual Activity; Consequences of Sex - HIV/STI; Consequences of Sex - Pregnancy; Managing Pressure to Engage in Sexual Activity through the Lens of Social Media; Financial Literacy; Careers; Post secondary Education; Wrap up and Close Out.
  The technology app will include curriculum support and additional resources.
  Students will have access to the mobile app after the in school programming ends. The intent is for students to have access to portions of the app that deal with self developed goals and progress monitoring for goals, and resource material. This is similar to a student having continued access to a textbook/other class materials.
  Interventions: Other: DREAMS Curriculum
- Non DREAMS (Active Comparator): The control group experience will include health curriculum already adopted by the school district. Continued services as usual. The control group schools, for the most part, lack any formal pregnancy prevention services. All schools claim that lessons developed by the teachers meet the Texas Essential Knowledge Standards (TEKS). No outside services are provided to students and school based services are limited. The services offered at the schools is predominately abstinence based. Students attending the schools would need to initiate any services that are available within the community. The control group will not have access to the DREAMS curriculum or the technology-based application to enhance the DREAMS curriculum. The technology-based application will be a closed, password protected, system during the research trial.
  Interventions: Other: DREAMS Curriculum

INTERVENTIONS:
Other: DREAMS Curriculum — Teen Pregnancy Prevention Curriculum as described in arm/group description.

SUMMARY:
The study is a an evaluation of the teen pregnancy prevention curriculum Decisions, Responsibility, Empowerment, Accountability, Motivations & Success (DREAMS) through a random control trial. The evaluation will take place in high schools in the greater Houston area. Five cohorts of two classes each in ten HS schools will be used. Randomization will occur each semester for five semesters. Curriculum is ten modules in length delivered in 45 minute classes twice a week for five weeks.

DETAILED DESCRIPTION:
The study is a an evaluation of the teen pregnancy prevention curriculum Decisions, Responsibility, Empowerment, Accountability, Motivations & Success (DREAMS) through a random control trial. The evaluation will take place in high schools in the greater Houston area. Five cohorts of two classes each in ten HS schools will be used. Randomization will occur each semester for five semesters. Curriculum is ten modules in length delivered in 45 minute classes twice a week for five weeks.

ELIGIBILITY:
Inclusion Criteria:

Age 13-19; enrolled in participating high school health class; passive consent received;

Exclusion Criteria:

Students who enrolled in classes post baseline. Students who had previously failed the HS course and was already exposed to DREAMS curriculum.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who had sex without a condom | immediately post-intervention, 6-months and 12-months-post intervention
  Number of participants who had sex without a condom. The relative difference of condom usage during penile-vaginal sex acts in the intervention versus control group at post-intervention, 6-months and 12-months post-intervention.
Number of participants who ever had sex | immediately post-intervention, 6-months and 12-months-post intervention
  Number of participants who ever had sex. The relative difference of ever having sex (penile-vaginal sex acts) in the intervention versus control group at post-intervention, 6-months and 12-months post-intervention.
Number of penile-vaginal sex acts | immediately post-intervention, 6-months and 12-months-post intervention
  Number of penile-vaginal sex acts. The relative difference of the number of penile-vaginal sex acts in the intervention versus control group at post-intervention, 6-months and 12-months post-intervention.
Number of participants who used other birth control methods | immediately post-intervention, 6-months and 12-months-post intervention
  Number of participants who used other birth control methods. The relative difference of birth control methods (e.g., the pill, the patch) during penile-vaginal sex acts in the intervention versus control group at post-intervention, 6-months and 12-months post-intervention.
Number of participants who had an STI | immediately post-intervention, 6-months and 12-months-post intervention
  Number of participants who had an STI. The relative difference of reported STI in the intervention versus control group at post-intervention, 6-months and 12-months post-intervention.
Number of participants who increased knowledge concerning risks associated with unprotected sex | immediately post intervention
  Number of participants who increased knowledge concerning risks associated with unprotected sex. The relative difference of knowledge gained in the intervention versus control group at immediately post-intervention.

SECONDARY OUTCOMES:
Number of participants (by gender, age, and race/ethnicity) who had had a teenage pregnancy | 12-months-post intervention
  Number of participants (by gender, age, and race/ethnicity) who had had a teenage pregnancy. The relative difference of teenage pregnancies (among genders, ages, and race/ethnicity) in the intervention versus control group at 12-months post-intervention.
Number of participants who had had a teenage pregnancy | 12-months-post intervention
  Number of participants who had had a teenage pregnancy. The relative difference of teenage pregnancies in the intervention versus control group at 12-months post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Bee Busy Inc., Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided